CLINICAL TRIAL: NCT00184327
Title: Change Across Intensive Inpatient Family Treatment in Child and Adolescent Psychiatry. A Multi-site Study of Parents and Children in Inpatient Family Treatment
Brief Title: Changes Following Inpatient Child-oriented Family Treatment
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Haukeland University Hospital (Other); St. Olavs Hospital (Other); Helse Nord-Trøndelag HF (Other); Namsos Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Forskpro p03000213
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Psychiatric Disorders
Keywords: Severe and longstanding psychiatric symptoms in children
MeSH Terms: conditions — Mental Disorders | interventions — Adolescent Psychiatry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Intensive family therapy - inpatient — 2-4 weeks (5days) family inpatient assessment and treatment
Behavioral: Diagnostic assessment - child and adolescent psychiatry

SUMMARY:
Children receiving IFT (intensive family therapy) were assessed for symptom profile and global functioning before admission, 3 months after discharge and 1 year after discharge. Children were assessed by parents, children, their teachers and themselves. Parents were assessed by themselves at the same points in time through psychological self-report questionnaires.

The study is intended to explore covariates to change in children as well as in parents during (pre-treatment) the treatment and follow-up periods.

DETAILED DESCRIPTION:
IFT is an intensive combinatory family treatment which is child-oriented, and traditionally used in an inpatient family treatment unit in child and adolescent psychiatry.

Measures include ones on bonding (PBI), personality traits (NEO-PI), anxiety and depressive symptoms (HADS), attributional tendencies (PAT) and social desirable responding (BIDR). A subgroup was also assessed before a waiting period (pre-treatment).

ELIGIBILITY:
Inclusion Criteria:

* Family offered inpatient family treatment in child and adolescent psychiatry.

Exclusion criteria

* inpatient treatment terminated prematurely

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Family offered inpatient family treatment in child and adolescent psychiatry
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2002-01; Primary Completion 2006-12 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tormod Rimehaug, Asst. Prof., Principal Investigator — Norwegian University of Science and Technology (NTNU), Faculty of Medicine, Dept. of Neuroscience, Center for Child and Adolescent Mental Health
Locations (5):
- Norway (5):
  - Haukeland University Hospital, Helse Bergen, Bergen
  - Levanger Hospital, Levanger
  - Namsos Hospital, Namsos
  - Norwegian University of Science and Technology (NTNU), Faculty of Medicine, Dept. of Neuroscience, Center for Child and Adolescent Mental Health, Trondheim
  - St.Olav Hospital, Trondheim

REFERENCES:
- [Result] Rimehaug T, Berg-Nielsen TS, Wallander J. Change in self-reported emotional distress and parenting among parents referred to inpatient child psychiatric family treatment. Nord J Psychiatry. 2012 Sep;66(4):260-7. doi: 10.3109/08039488.2011.630752. Epub 2011 Nov 16. PMID 22087555